CLINICAL TRIAL: NCT00500019
Title: Uterine Flora During Elective and Urgent Cesarean Sections and Its Relationship to Postpartum Complications.
Brief Title: Uterine Flora During Elective and Urgent Cesarean Sections
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Professor Jacob Bornstein, Department Obstetrics & Gynecology, Western Galilee Hospital, Nahariya, Israel
Other Study IDs: 1-Bornstein
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Endometritis
MeSH Terms: conditions — Endometritis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Uterine bacteriological cultures
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1.: Elective Cesarean sections
- 2.: Non-elective cesarean section

SUMMARY:
Hypothesis: The bacterial flora of the uterus during elective Cesarean sections differs from the uterine flora during non-elective Cesarean sections. We want to study whether the uterine flora can predict post-cesarean febrile morbidity and endometritis.

DETAILED DESCRIPTION:
Objective: To evaluate the uterine flora at the time of elective and non-elective cesarean sections and to study the relationship to the development of postpartum fever and/or endometritis.

Methods: Eight-hundred women who will be delivered by cesarean section will be enrolled in this study. Cultures will be obtained during the surgery from the open uterine cavity after removal of the placenta. Data regarding postpartum morbidity would be collected.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery

Exclusion Criteria:

* Vaginal delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing cesarean sections in Western galilee Hospital
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2005-01; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To compare bacteriological growth between elective and non-elective cesarean section | 5 years

SECONDARY OUTCOMES:
To study the various bacteria growth in the uteri, and to compare type of bacteria to post-op morbidity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ido Solt, MD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Western Galilee Hospital, Nahariya, Israel